CLINICAL TRIAL: NCT04776096
Title: PHASE IV, MULTICENTRIC, DOUBLE-BLIND, RANDOMIZED, CONTROLLED,60 DAYS, PARALLEL GROUPS, SUPERIORITY STUDY, TO COMPARE THE EFFECTIVENESS AND TOXICITY OF BEPOTASTINE 1.5% PF vs. OLOPATADINE 0.2% WITH BAK IN TREATMENT OF ALLERGIC CONJUNCTIVITIS
Brief Title: Efficacy and Toxicity of Bepotastine 1,5% PF vs Olopatadine 0,2% With BAK on Allergic Conjunctivitis Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratorios Poen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANTILERG001-19
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — bepotastine besilate; Olopatadine Hydrochloride

STUDY DESIGN:
Intervention Model Description: MULTICENTRIC, DOUBLE BLIND, RANDOMIZED, CONTROLLED, 60 DAYS, GROUP PARALLEL GROUPS, TO SHOW SUPERIORITY.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bepotastine besilate 1,5% preservative free (Experimental): Bepotastine besilate 1,5% in preservative-free bottle, administered once a day during the morning.
  Interventions: Drug: Bepotastine Besilate 1.5% PF
- Olopatadine hydrochloride 0,2% with BAK (Active Comparator): Olopatadine hydrochloride 0,2% with BAK as preservative, administered once a day during the morning.
  Interventions: Drug: Olopatadine Hydrochloride 0.2% BAK

INTERVENTIONS:
Drug: Bepotastine Besilate 1.5% PF — Bepotastine besilate 1,5% Preservative free ophthalmic solution
  Other Names: TRALER LC
  Arms: Bepotastine besilate 1,5% preservative free
Drug: Olopatadine Hydrochloride 0.2% BAK — Olopatadine hydrochloride 0.2% with BAK as preservative
  Arms: Olopatadine hydrochloride 0,2% with BAK

SUMMARY:
The present study will be carried out to evaluate the antiallergic efficacy of Bepotastine besilate 1.5% free of preservatives versus standard treatment with 0.2% Olopatadine hydrochloride with 0.1% benzalkonium chloride as preservative in adult patients diagnosed with allergic conjunctivitis.

The antiallergic efficacy will be evaluated by the reduction of ocular signs and symptoms and by the resolution of non-ocular symptoms (rhinorrhea, congestion, and nasal pruritus), as well as the effect of the preservative and its relationship with the cytotoxicity of the ocular surface. Also will evaluate the safety of both products.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old.
* Clinical diagnosis of allergic conjunctivitis and active allergy with at least 2 points on itching and hyperemia scale.
* Patients with history of allergic conjunctivitis.
* Patients who accept no to wear contact lens during the duration of the trial.
* Patients who accept no to use any other medication by any delivery route.
* Patients with intraocular pressure controlled (less than 18 mmhg)

Exclusion Criteria:

* Patients who have undergone refractive surgery within the 6 months prior to the start of the study
* Patient with ocular or systemic active diseases
* Patients who are participating in another trial
* Patients who have used eye medication in the last 15 days and/or who have received anti-inflammatory drugs (corticosteroids and/or NSAIDs) and/or antihistamines by mouth or intravenous.
* Patients hypersensitive to any component of the products: Bepotastine besilate, sodium chloride, monosodium phosphate dihydrate, sodium hydroxide, Olopatadine hydrochloride, benzalkonium chloride, dibasic sodium phosphate, hydrochloric acid, edetate disodium or povidone K29 / 32.
* Women who are breastfeeding and pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
Ocular itching | Baseline, Day 15, Day 30, Day 45, Day 60
  Change of 1 point of scale 0-3 (none, mild, moderate, severe) in at least 1 visit between gruops.

SECONDARY OUTCOMES:
Eye burning | Baseline, Day 15, Day 30, Day 45, Day 60
  Differences between treatments. Scale 0-3 (none, mild, moderate, severe)
Eye lacrimation | Baseline, Day 15, Day 30, Day 45, Day 60
  Differences between treatments. Scale 0-3 (none, mild, moderate, severe)
Foreign body sensation | Baseline, Day 15, Day 30, Day 45, Day 60
  Differences between treatments. Scale 0-3 (none, mild, moderate, severe)
Rhinorrhea | Baseline, Day 15, Day 30, Day 45, Day 60
  Differences between treatments. Scale 0-3 (none, mild, moderate, severe)
Nasal congestion | Baseline, Day 15, Day 30, Day 45, Day 60
  Differences between treatments. Scale 0-3 (none, mild, moderate, severe)
Nasal pruritus | Baseline, Day 15, Day 30, Day 45, Day 60
  Differences between treatments. Scale 0-3 (none, mild, moderate, severe)
Eyelid swelling | Baseline, Day 15, Day 30, Day 45, Day 60
  Differences between treatments. Scale 0-3 (none, mild, moderate, severe)
Visual Acuity | Baseline and Day 60
  Improve from baseline.
Meniscus height | Baseline, Day 15, Day 30, Day 45, Day 60
  Differences between treatments.
Conjunctival hyperemia | Baseline, Day 15, Day 30, Day 45, Day 60
  Differences between treatments. Scale 0-3 (none, mild, moderate, severe)
Chemosis | Baseline, Day 15, Day 30, Day 45, Day 60
  Differences between treatments. Scale 0-3 (none, mild, moderate, severe)
Eye discharge | Baseline, Day 15, Day 30, Day 45, Day 60
  Differences between treatments. Scale 0-3 (none, mild, moderate, severe)
Conjuctival impression cytology | Baseline, Day 30, Day 60
  Differences between treatments. Nelson classification.
Adverse reactions | Baseline, Day 15, Day 30, Day 45, Day 60.

CONTACTS AND LOCATIONS:
Locations (4):
- Argentina (4):
  - Hospital de Alta Complejidad El Cruce - Nestor Kirchner, CABA
  - Hospital Santa Lucía, CABA
  - Instituto Oftalmológico Pedro Lagleyze, CABA
  - Hospital Churruca - Visca, CABA

IPD SHARING:
Plan to Share IPD: Undecided